CLINICAL TRIAL: NCT02613299
Title: Surgery for Mesothelioma After Radiation Therapy "SMART" for Resectable Malignant Pleural Mesothelioma
Status: Terminated | Type: Observational
Why Stopped: slow accrual related to change in standard-of-care treatment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Dennis Wigle, Principal Investigator, Mayo Clinic
Other Study IDs: 15-007644
Record Dates: First submitted 2015-11-20; First posted 2015-11-24 (Estimated); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Mesothelioma; Solitary Fibrous Tumor of the Pleura
MeSH Terms: conditions — Mesothelioma; Solitary Fibrous Tumor, Pleural

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The purpose of this study is to determine whether radiation therapy decreases tumor size and tumor spread. The investigators will consent subjects that have been diagnosed with mesothelioma and will undergo radiation therapy followed by surgical resection as their standard of care. The investigators will collect data from past and future medical records as well as data regarding their health status for their lifetime by reviewing life status, treatment status and CT scans.

ELIGIBILITY:
Inclusion Criteria:

* Subject provides informed consent
* Subject is >18 years of age
* Subject is deemed competent for making medical decisions
* Subject is scheduled to undergo radiation followed by extrapleural pneumonectomy.
* Subject is a surgical candidate
* A negative pregnancy test is required in women of child-bearing potential, as standard of care.

Exclusion Criteria:

* Subject is <18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving treatment at the Mayo Clinic Rochester that have been diagnosed with mesothelioma and will undergo radiation therapy followed by surgical resection as their standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2016-06-14 (Actual); Primary Completion 2025-05-29 (Actual); Study Completion 2025-05-29 (Actual)

PRIMARY OUTCOMES:
Survival status upon review of patient records annually | Up to 10 years

CONTACTS AND LOCATIONS:
Overall Officials: Dennis Wigle, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials